CLINICAL TRIAL: NCT03381417
Title: A Randomized, Double-blind, Parallel Study Comparing Efficacy and Safety of Pegcyte (Nanogen) and Reference Product Neulastim (Roche) for Prevention of Chemotherapy (Accelerated AC Regimen)Induced Neutropenia in Breast-cancer Patients.
Brief Title: Nanogen Pegcyte Clinical Study for the Prevention of CIN in Breast-cancer Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanogen Pharmaceutical Biotechnology Joint Stock Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NNG05
Record Dates: First submitted 2017-12-11; First posted 2017-12-22 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pegcyte (Nanogen pegfilgrastim) (Experimental): 6 mg in each cycle
  Interventions: Drug: pegcyte
- Neulastim (Roche pegfilgrastim) (Active Comparator): 6 mg in each cycle
  Interventions: Drug: Neulastim

INTERVENTIONS:
Drug: pegcyte — Eligible patients are scheduled to receive three cycles of chemotherapy every two weeks. During each chemotherapy cycle pegfilgrastim is injected s.c. post chemotherapy application.
  Other Names: pegfilgrastim
  Arms: Pegcyte (Nanogen pegfilgrastim)
Drug: Neulastim — Eligible patients are scheduled to receive three cycles of chemotherapy every two weeks. During each chemotherapy cycle pegfilgrastim is injected s.c. post chemotherapy application.
  Other Names: pegfilgrastim
  Arms: Neulastim (Roche pegfilgrastim)

SUMMARY:
Accelerated AC regimen-Doxorubicin 60 mg/m2,Cyclophosphamide 600 mg/m2 on day 1 & day 14 of each cycle along with G-CSF support for up to 4 cycles, followed by Paclitaxel 175 mg/m2 in the next 4 cycles is the standard clinical practice in Vietnam for breast cancer, this regimen is to facilitate the dose-dense schedule, patients receive every-2-week therapy along with G-CSF support. the accelerated dose-dense schedule improve disease-free and overall survival among women with breast cancer .Primary objective of this study is to compare the efficacy and safety of Nanogen's Pegcyte and Roche's Neulastim for prevention of chemotherapy (Accelerated AC regimen)-induced neutropenia on breast cancer patients. Breast cancer patients scheduled to receive myelosuppressive chemotherapy (AC regimen) will be recruited in this trial. All eligible patients receive single subcutaneous injection of study drugs 24 hours after chemotherapy administration in each cycle for 3 consecutive cycles. Efficacy and safety assessments will be assessed based on the incidence of severe neutropenia in combination of temperature > 38.3℃ or sepsis or life threatening infection and incidence of serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 - 65 years.
* Patients with histological confirmed primary invasive breast cancer; stage I, II or III.
* Patients had no prior chemotherapy treatments.
* Patients scheduled to undergo myelosuppressive Doxorubicin and Cyclophosphamide chemotherapy for 04 cycles, and Paclitaxel chemotherapy for the next 04 cycles; patients were available for 14 days of each cycle for the first 03 chemotherapy cycles.
* Patients with baseline ANC ≥ 1.5 x 109/L, PLT ≥ 100 x 109/L, HgB ≥ 9 g/dL, WBC ≥ 3,000/mL and albumin ≥ 3.0 g/dL.
* Performance status as per ECOG (Eastern Cooperative Oncology Group) score 0, 1 or 2.
* Willing to give written and signed informed consent.

Exclusion Criteria:

* Patients with prior exposure of G-CSF or GM-CSF or its pegylated products in clinical development less than 6 months prior to randomization.
* Myelotoxic concomitant treatment such as chloramphenicol, methotrexate, immunomodulating agents, interferons during 10 days before randomization.
* Received systemic antibiotic treatment within 72 hours of chemotherapy.
* Chronic use of corticosteroids, prior bone marrow or stem cell transplant.
* Patients who had an immediate/ concurrent exposure to radiotherapy or surgery (within 4 weeks).
* Severe medical disease: cardiovascular, hepatic, renal, pulmonary…
* Known cases of hematological disease (sickle cell anemia, AML…)
* History of HIV positive, active hepatitis.
* Pregnant and lactating women or patients planning to become pregnant.
* Known allergic reactions to study medications.
* Positive to anti-pegfilgrastim antibody test

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — breast cancer
Enrollment: 128 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who developed Febrile neutropenia in cycle 1,2 and 3 | 0 to 42 days)

SECONDARY OUTCOMES:
Incidence of grade 4 severe neutropenia | in cycle 1,2 and 3 (0 to 14 , 28 and 42 days)
Incidence of antibiotics use | in cycle 1,2 and 3 (0 to 14 , 28 and 42 days)
Incidence of adverse events | in cycle 1,2 and 3 (0 to 14 , 28 and 42 days)
Changes in laboratory safety parameters | in cycle 1,2 and 3 (0 to 14 , 28 and 42 days)
  including vital signs
Presence of antibodies against Pegfilgrastim | at the end of cycle 3 (42 day)

CONTACTS AND LOCATIONS:
Locations (1):
- Vietnam National Cancer Institute (Hospital K), Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided